CLINICAL TRIAL: NCT01257867
Title: Lithia Water Study: Effects of Lithia Water on BDNF and Oxidative Stress Markers in Healthy Male Participants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated by the Principal Investigator
Sponsor: University of British Columbia (Other)
Collaborators: Aquaceutica Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H10-03015
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Oxidative Stress
Keywords: Brain-derived neurotrophic factor; Oxidative stress; Neurogenesis; Lithium; Lithia water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lithia spring water (Experimental): Lithia water (active) for 4 weeks then placebo water for 4 weeks
  Interventions: Dietary Supplement: Lithia water
- Natural spring water (Placebo Comparator): Placebo water for 4 weeks then lithia water (active) for 4 weeks
  Interventions: Dietary Supplement: Natural spring water with negligible lithium levels

INTERVENTIONS:
Dietary Supplement: Lithia water — Oral intake of approximately 2 litres (2L) daily for 4 weeks
  Other Names: EDJ lithia spring water; (previous) Ilumati lithia spring water
  Arms: Lithia spring water
Dietary Supplement: Natural spring water with negligible lithium levels — Oral intake of approximately 2 litres (2L) daily for 4 weeks
  Arms: Natural spring water

SUMMARY:
This study investigates the effects of daily use of lithia water on blood tests of neuronal oxidative stress, mood, and well-being. Lithia water is a type of pure spring water containing trace levels of lithium, which is a naturally occurring mineral. Neuronal oxidative stress is caused by normal chemical reactions in the human body that sometimes result in damage to brain cells. Participation in this study will last for 8 weeks and includes daily use of study water for drinking.

The primary objective of this pilot study is to test the hypothesis that, in healthy male participants, daily use of lithia water will improve neurogenesis and antioxidant capacity as measured by serum levels of brain-derived neurotrophic factor (BDNF) and oxidative stress markers. Secondary objectives will include examining self-reported changes in mood, cognition, and well-being.

DETAILED DESCRIPTION:
There is some indication from epidemiological studies that areas with trace concentrations of lithium in drinking water have lower rates of suicide. This study will evaluate the effects of drinking EDJ (pronounced "edge") lithia spring water (which comes from a natural spring in the Rocky Mountains and contains trace amounts [0.68 mg/litre] of lithium) for 4 weeks, compared to drinking commercially available bottled water (which contains no lithium at all) for 4 weeks.

This pilot study has been designed as an 8-week randomized, counterbalanced, crossover study in 15 healthy male participants. Eligible participants will use lithia water or control water for daily ingestion for 4 weeks, then cross over to the other condition for another 4 weeks. At baseline and after each 4-week condition, participants will complete self-report questionnaires of mood, cognition and well-being, and blood samples will be assayed for BDNF and oxidative stress protein markers.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 19-35 years. [Note: women are excluded in this pilot study because the variable effects of female sex hormones on oxidative stress markers and neurogenesis];
* No current, past or family history (in first-degree relatives) of a major psychiatric disorder or alcohol/substance abuse/dependence;
* Non-smokers [because smoking is associated with increased oxidative stress];
* No active medical condition (e.g., thyroid disease);
* No regular use of prescribed or over-the-counter medications or illicit substances;
* Negative urine drug-screening test; and
* Competency to give informed consent.

Exclusion Criteria:

* See above

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in BDNF levels at 4 weeks | Baseline, Wk 4, Wk 8
  Blood samples will be assayed for brain-derived neurotrophic factor

SECONDARY OUTCOMES:
Standardized, validated questionnaires querying mood and quality of life | Baseline, Wk 4, Wk 8
Standardized, validated questionnaires regarding cognitive functioning | Baseline, Wk 4, Wk 8
Change from Baseline in oxidative stress protein markers at 4 weeks | Baseline, Wk 4, Wk 8
  Blood samples will be assayed for oxidative stress protein markers (superoxide dismutase, catalase, glutathione peroxidase, and TBARS)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W Lam, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Department of Psychiatry, Vancouver, British Columbia, Canada

REFERENCES:
- See also: University of British Columbia — http://www.ubc.ca